CLINICAL TRIAL: NCT06577155
Title: The Effect of Nalbuphine as an Adjuvant to Levobupivacaine in Subarachnoid Anesthesia in Total Hip Arthroplasty. A Double-blind, Randomized, Controlled Study.
Brief Title: Spinal Nalbuphine for Analgesia in Total Hip Arthroplasty
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Collaborators: Anastasios Mpontozis (Unknown)
Responsible Party: Principal Investigator, Alexandros Makris, Consultant Anaesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10542/22-05-2024
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Total Hip Arthroplasty; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Levobupivacaine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E (Active Comparator): Spinal levobupivacaine
  Interventions: Drug: Levobupivacaine
- N (Active Comparator): Spinal levobupivacaine plus nalbuphine
  Interventions: Drug: Levobupivacaine plus nalbuphine

INTERVENTIONS:
Drug: Levobupivacaine — Regional anesthesia / analgesia
  Arms: E
Drug: Levobupivacaine plus nalbuphine — Regional anesthesia / analgesia
  Arms: N

SUMMARY:
60 patients ASA I-III, undergoing total hip arthroplasty were randomly assigned, into one of two groups, namely group E (n=30), where levobupivacaine will be administeral intrathecally ; and group N (n=30), where levobupivacaine plus nalbuphine will be administeral intrathecally. All patients will receive a standardized multimodal analgesic regimen, including a PENG block and PCA morphine. Morphine consumption during the first 24 hours postoperatively will be measured and additionally the investigators will record: Time of morphine first dose administration, NRS scores in static and dynamic conditions in 4 hours, 6 hours, 12 hours, 18 hours, 24 hours, 36 hours and 48 hours postoperatively, complications, patient satisfaction and duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-III
* Patients scheduled for total hip arthroplasty

Exclusion Criteria:

* BMI above 40
* Serious psychiatric, mental and cognitive disorders
* Contraindication for central and/or peripheral nervous blockade
* History of allergic or other adverse reactions on the agents used in the study
* Chronic opioid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours
NRS scores | 48 hours

SECONDARY OUTCOMES:
sensory block level | 1 hour
motor block level | 1 hour
sensory block onset | 1 hour
motor block onset | 1 hour
sensory block duration | 4 hours
motor block duration | 4 hours
Complications | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Ελλάδα (+30), Greece

IPD SHARING:
Plan to Share IPD: No